CLINICAL TRIAL: NCT06754033
Title: Comparison of Ganglion Impar Block With Physical Therapy Versus Caudal Epidural Steroid Injection With Physical Therapy for Patients With Coccydynia
Brief Title: Ganglion Impar Block With Physical Therapy vs Caudal Epidural Steroid Injection With PT for Patients With Coccydynia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/766
Record Dates: First submitted 2024-12-13; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Coccyx Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Diagnostic Test: Interventional group I
- Interventional group II (Active Comparator)
  Interventions: Combination Product: Interventional group II

INTERVENTIONS:
Diagnostic Test: Interventional group I — Intervention Details: Participants in this arm will receive a Ganglion Impar Block, a minimally invasive injection aimed at blocking pain signals from the coccyx region (Ganglion Impar Block using Triamcinolone Acetate (40 mg) and Bupivacaine (0.25%) administered with a 22G Spinal Needle under Fluoroscopic Guidance). Participants in this arm will receive a Ganglion Impar Block, a minimally invasive procedure involving the administration of Triamcinolone Acetate (a corticosteroid) and Bupivacaine (a local anesthetic). This is intended to block pain signals originating from the coccyx region. The procedure will be conducted under fluoroscopic guidance to ensure precise delivery. The injection will be complemented by a structured physical therapy program, including heat therapy, ultrasound, posture training, core strengthening exercises, and mobility activities to improve pain relief and functional capacity.
  Arms: Interventional group I
Combination Product: Interventional group II — Intervention Details: Participants in this arm will receive a Caudal Epidural Steroid Injection Caudal Epidural Steroid Injection using Triamcinolone Acetate (40 mg), Bupivacaine (0.25%), and Normal Saline (6 mL) administered with a 22G Spinal Needle under Fluoroscopic Guidance), designed to deliver anti-inflammatory medication directly to the epidural space, thereby reducing inflammation and pain. This will also be paired with a tailored physical therapy program, focusing on similar modalities as in Arm 1, including heat therapy, ultrasound, posture training, and strengthening exercises. The objective is to enhance pain relief and functional recovery in the context of coccydynia.
  Arms: Interventional group II

SUMMARY:
The study aims to evaluate the efficacy of two treatment modalities for patients suffering from coccydynia: Ganglion Impar Block (GIB) combined with physical therapy, and Caudal Epidural Steroid Injection (CESI) also accompanied by physical therapy. Coccydynia, characterized by pain in the coccygeal region, can significantly impair daily functioning and quality of life.

DETAILED DESCRIPTION:
Participants were assessed using various outcome measures, including the SF-12, Oswestry Disability Index (ODI), and Numeric Pain Rating Scale (NPRS). Data collection will occur at baseline and through four follow-up points over 16 weeks, allowing for a comprehensive evaluation of both immediate and long-term treatment effects. By comparing these two interventions, the study seeks to determine which approach yields superior results in alleviating pain and improving functional outcomes for patients with coccydynia, thereby contributing valuable insights into the management of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with age 18-65 diagnosed with chronic coccydynia for at least 3 months were recruited.
* Participants who will be willing & able to adhere to the study protocol.
* Including participants who will be attending follow-up appointments & completing outcome measures.
* Participants who will be able to understand & provide written informed consent.
* Participants with a complete screening of other medical conditions and previous medical records.

Exclusion Criteria:

* Participants with previous surgery on the coccyx or lumbosacral spine, pregnancy or breastfeeding, history of bleeding disorders or anticoagulant use, active infection, or significant medical condition that could pose a safety risk during the procedures (GIB or CESI) was omitted.
* Patients above the age of 65 were eliminated to reduce confounding by age-related health concerns and to provide a more homogenous study population for more accurate treatment outcomes.
* Participants with neurological conditions affecting pain perception or sensation were excluded.
* Participants with known allergies to medications used in the study (local anesthetic, steroid for injections) were not part of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 12 Months
  Used as the primary outcome measure. Participants will rate their pain intensity on a scale of 0 to 10, with 0 indicating no pain and 10 indicating the worst possible pain. This measure will assess changes in pain levels from baseline through various follow-up points.
Oswestry Disability Index (ODI) | 12 months
  The Oswestry Disability Index will serve as the secondary outcome measure. This questionnaire evaluates the degree of disability experienced by participants due to their pain, focusing on various aspects of daily living and functional capacity. Additionally, the SF-12 health survey will be used to measure the overall health-related quality of life, providing further insights into the impact of the interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghurkee Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No